CLINICAL TRIAL: NCT03329430
Title: Influence of Custom Foot Orthoses on Venous Status
Brief Title: Custom Foot Orthoses & Venous Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, PhD, MSc, PT, Universidad de León
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: foot_orthoses_venous_status
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Foot; Foot Orthoses; Photoplethysmography; Venous Stasis
MeSH Terms: conditions — Varicose Ulcer | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foot orthoses (Experimental): Customize foot orthoses
  Interventions: Other: Foot orthoses

INTERVENTIONS:
Other: Foot orthoses — Customized foot orthoses

SUMMARY:
The purpose of the research is to compare the influence of customized foot orthoses use on the venous status among healthy female and male subjects. This is a quasi-experimental study which included 20 healthy subjects. Sociodemographic and medical record data are registered. Furthermore,venous function is evaluated by plethysmography, first, without orthoses and, after 20 days, with orthoses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects.

Exclusion Criteria:

* Prior diagnosed conditions such as neurological, vascular or traumatic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Venous filling time | Change from Baseline venous filling time at 1 month
  Seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde do Vale do Ave, Vila Nova de Famalicão, Vila Nova de FamalicÃ£o, Portugal

IPD SHARING:
Plan to Share IPD: No